CLINICAL TRIAL: NCT06859983
Title: The Effect of Progressive Muscle Relaxation Exercises on Fatigue Severity and Sleep Quality in Emergency Department Nurses: A Self-Controlled Quasi-Experimental Study
Brief Title: The Effect of Progressive Muscle Relaxation Exercises on Fatigue Severity and Sleep Quality in Emergency Department Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Sumeyye Akcoban, Lecturer, Mustafa Kemal University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HMKU-KMY-SA-04
Record Dates: First submitted 2025-02-28; First posted 2025-03-05 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-02

CONDITIONS: Progressive Muscle Relaxation Exercise
Keywords: Progressive muscle relaxation exercise; Emergency department; nurse; fatigue severity; sleep quality
MeSH Terms: conditions — Emergencies; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Emergency department nurses (Experimental): In the first phase, data collection will begin on the first day (n=35) with nurses, and the nurse introductory information form will be collected through face-to-face interviews. Then, at the end of each week during the 4-week period, nurses will complete the "Fatigue Severity Scale" and the "Pittsburgh Sleep Quality Index (PSQI)" four times. This will complete the pre-intervention evaluation.
  Interventions: Behavioral: progressive relaxation exercise

INTERVENTIONS:
Behavioral: progressive relaxation exercise — he researcher will provide approximately 45 minutes of information about relaxation exercises to the nurses. During the application of progressive relaxation exercises, the necessary precautions to be taken during and after the exercise will be explained to the nurses. In the study, a sound recording that includes the PRE will be uploaded to each nurse's phone. The relaxation exercises CD created by the Turkish Psychologists Association will be used for the sound recording. The first section of the CD, which is 10 minutes long, defines deep relaxation, its purpose, and the precautions to be taken during the exercise. The second 30-minute section explains the relaxation exercises with the sound of a stream and verbal instructions. The third 30-minute section contains only relaxation music without any verbal instructions. After the training, nurses will be given the sound recording in CD form. Nurses will be asked to perform the PRE according to the instructions. They will be instructed

SUMMARY:
Emergency departments are critical units where patients with life-threatening conditions and acute illnesses receive rapid interventions. Nurses working in these units aim to provide the best possible healthcare by intervening with patients at high risk of life-threatening situations. However, long working hours, inadequate working conditions, high stress, and critical patient care often lead to physiological issues among nurses. Fatigue and insomnia, which are commonly linked to burnout, are among the most frequent physiological problems.

Insomnia is a condition characterized by poor and irregular sleep patterns occurring within a 24-hour period due to disruption of the circadian rhythm. Chronic insomnia, if persistent, triggers fatigue. Fatigue is a subjective condition that, when prolonged, negatively affects nurses' daily activities and reduces job performance. Moreover, increasing fatigue has significant adverse effects on alertness, attention, judgment, and mood. These effects can lead to accidents, errors in practice, and injuries.

DETAILED DESCRIPTION:
Progressive relaxation exercises reduce blood levels of epinephrine and norepinephrine, oxygen consumption, blood pressure, metabolic rate, heart rate, muscle tension, lactic acid levels, pain and fatigue. On the other hand, concentration increases endorphin release, reduces insomnia and provides mental well-being. When the literature was examined, progressive relaxation exercise practices were performed on patients with rheumatoid arthritis and it was determined that there were positive effects on insomnia and fatigue levels in patients at the end of a six-week period. In another study evaluating the effectiveness of progressive relaxation exercise in dialysis patients, it was found that the fatigue level of the patients decreased. Again, when the literature was examined, two studies evaluating the effectiveness of progressive relaxation exercise on intensive care nurses were found in our country. In these studies conducted with intensive care nurses, it was reported that progressive relaxation exercises had a positive effect on fatigue.

In line with our research, no study was found to examine the effect of progressive relaxation exercises applied to nurses working in the emergency department on fatigue severity and sleep quality.

Translated with www.DeepL.com/Translator (free version)

ELIGIBILITY:
Inclusion Criteria:

* Working in the emergency service unit,
* No psychiatric disorder,
* Can do progressive relaxation exercises,
* Apply progressive relaxation exercises for one month,
* No disease that prevents progressive relaxation exercise,

Exclusion Criteria:

* Nurses who do not meet the inclusion criteria will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-03-08 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Nurse Introductory Information Form | he necessary evaluation will be made at the end of the first week.
  The data collection form consists of 12 statements developed by the researchers as a result of the literature review, questioning age, gender, educational status, marital status, working time in the profession, working style, sleep quality and fatigue.
Fatigue Severity Scale | The necessary evaluation will be made at the end of the first week.
  The scale developed by Krup (1989) consists of nine items assessing the general effect of fatigue on daily activities. The Turkish validity and reliability of the scale was performed by Armutlu et al. In the scale, individuals are asked to rate the fatigue they felt during the past week from 1 to 7. Each section is scored between 1 (strongly disagree) and 7 (strongly agree) (add 2 to 6). The total score is calculated by averaging the nine items. The cut-off value for pathological fatigue is set at 4 and above. The lower the total score, the lower the fatigue. Cronbach's alpha coefficient of the scale was 0.94 in the study of Armutlu et al.
Pittsburgh Sleep Quality Index | The necessary evaluation will be made at the end of the first week.
  expressed in a single item, while others are expressed in a group of several items. Each item score ranges from "0" to "3". The total PDQI score is between 0 and 21. A score above 5 indicates that the sleep quality of the individual is poor. The Cronbach alpha value of the scale was found to be 0.80 in the study of Ağargün et al.

SECONDARY OUTCOMES:
Nurse Introductory Information Form | The necessary evaluation will be made at the end of the first week.
  The data collection form consists of 12 statements developed by the researchers as a result of the literature review, questioning age, gender, educational status, marital status, working time in the profession, working style, sleep quality and fatigue.
Fatigue Severity Scale | The necessary evaluation will be made at the end of the second week.
  The scale developed by Krup (1989) consists of nine items assessing the general effect of fatigue on daily activities. The Turkish validity and reliability of the scale was performed by Armutlu et al. In the scale, individuals are asked to rate the fatigue they felt during the past week from 1 to 7. Each section is scored between 1 (strongly disagree) and 7 (strongly agree) (add 2 to 6). The total score is calculated by averaging the nine items. The cut-off value for pathological fatigue is set at 4 and above. The lower the total score, the lower the fatigue. Cronbach's alpha coefficient of the scale was 0.94 in the study of Armutlu et al.
Pittsburgh Sleep Quality Index | The necessary evaluation will be made at the end of the second week.
  The scale developed by Krup (1989) consists of nine items assessing the general effect of fatigue on daily activities. The Turkish validity and reliability of the scale was performed by Armutlu et al. In the scale, individuals are asked to rate the fatigue they felt during the past week from 1 to 7. Each section is scored between 1 (strongly disagree) and 7 (strongly agree) (add 2 to 6). The total score is calculated by averaging the nine items. The cut-off value for pathological fatigue is set at 4 and above. The lower the total score, the lower the fatigue. Cronbach's alpha coefficient of the scale was 0.94 in the study of Armutlu et al.

CONTACTS AND LOCATIONS:
Locations (1):
- Hatay Mustafa Kemal University, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No